CLINICAL TRIAL: NCT06910085
Title: Kettlebell-classroom: Feasibility and Effect of a Daily Dose of Resistance Training in Primary School Children - a Control\ed Trial
Brief Title: Kettlebell-classroom Training
Acronym: kettleclass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-01074; 2024-01074 (Other: ethics committee)
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Schools; Primary Health Care; Resistance Training; Muscle Strength; Feasibility Studies; Schools / Organization & Administration; Preventive Health Services
Keywords: Kettlebell Training; Daily school routine; Teacher involvement; Primary school; Physical education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kettlebell training (Active Comparator): The intervention involves daily, supervised resistance training sessions for primary school children, integrated directly into the classroom setting. Over a period of 7 weeks, participating second-grade school classes perform 15-minute kettlebell-based workouts every school day, totaling 35 sessions.
  The sessions are designed to be:
  Playful and age-appropriate
  Focused on whole-body strength and motor skill development
  Based on functional, multi-joint movements using bodyweight and kettlebells
  Adaptable to individual ability levels
  Including elements of teamwork and cooperation to enhance motivation and enjoyment
  The goal is to improve muscular strength, coordination, fitness, and psychosocial well-being, particularly in children from lower socio-economic backgrounds.
  Interventions: Behavioral: kettlebell-training
- regular schedule - control (No Intervention): The control group consists of parallel second-grade school classes that do not receive any active intervention during the study period. These students continue with their regular school routine and standard physical education classes, without the additional kettlebell training sessions.
  Like the intervention group, they:
  Undergo the same pre- and post-intervention test battery assessing strength, coordination, fitness, and anthropometric measures
  Are assessed during school hours using identical equipment and protocols
  Serve as a baseline comparator to evaluate the effectiveness and feasibility of the resistance training intervention

INTERVENTIONS:
Behavioral: kettlebell-training — 15 min of body weight or kettlebell loaded strength training
  Arms: kettlebell training

SUMMARY:
Physical fitness is a crucial health marker, predicting both cardiovascular and all-cause mortality. Muscular strength, an essential component of physical fitness, underpins physical and psychological well-being, particularly from childhood. Increasing sedentary behavior has led to rising obesity and cardiovascular disease rates in children, exacerbated by the COVID-19 pandemic and the emergence of pediatric dynapenia. Muscular fitness positively affects body composition, bone health, psychological health, and academic performance, and is necessary for fundamental motor skills.

In Basel, a ten-year trend shows declining physical fitness and rising obesity among primary school children, especially those from lower socio-economic backgrounds with less access to sports. This presents an opportunity to promote physical activity in schools. The "Kettlebell Classroom" project aims to introduce daily, playful resistance training with kettlebells over seven weeks in various schools, focusing on culturally and socially less integrated children.

Evidence supports the benefits of resistance training (RT) for children, including increased joint stability, improved motor skills, reduced injury risks, and increased spontaneous physical activity. Despite WHO recommendations for muscle and bone-strengthening activities three times a week, these guidelines are often unmet. This project aims to demonstrate the effectiveness of short, intensive exercise sessions for children, with the goal of expanding the initiative across Basel to improve health outcomes for all children.

DETAILED DESCRIPTION:
Study intervention The intervention emphasizes full-body exercises which are performed with the own body weight and kettlebells. On every weekday, the intervention classes will receive 15 min of supervised training over 7 weeks. This results in a total number of training sessions of 35 sessions. The movements and exercises in all phases are based on functional, multi-joint movements. The focus will be on age-appropriate whole-body strength and motor skill development. It will be designed with different, varying exercises, which can be individually tailored and adapted to the children's ability. Tailored to the group, the sessions will also include parts which engage social cooperation and teamwork, so that the children will experience a sense of competence, self-determination and enjoyment of exercise while enhancing motor skills and athletic ability.

ELIGIBILITY:
Inclusion Criteria:

* all of the selected second-graders who can participate in physical education lessons will be included in the study

Exclusion Criteria:

* Children with a medical certificate, that prohibits physical activity, will be excluded from performance testing and training intervention.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Maximal strength | seven week intervention
  The mid-thigh pull is measured on the force plate, as is the hand grip force (Leonardo Mechanograph® Novotec Medical GmbH, Pforzheim, Germany). The mid-thigh pull corresponds to a static deadlift, i.e. pulling up a bar in the centre of the thigh, and thus provides an image of the force transmission of the muscle loops up to the hand force to transfer the force to the measuring device. The test subject has a hip and knee angle of 135-140° and tries to pull as quickly and strongly as possible on the vertically fixed bar in the centre of the thigh. As the test subject is standing on the force plate, the transmitted force is measured precisely. In contrast to the dynamic 1-repetition maximum, this simple test offers a high level of safety as an isometric measurement and, in particular, has a high test-retest reliability. This measurement is therefore not only attractive to perform, but also makes it easy to analyse strength curves and maximum strength.

SECONDARY OUTCOMES:
Handgrip strength | seven week intervention
  The handgrip force is measured using a size-adjustable application to take into account the span of the respective hand size. The measurement is performed with the arm extended vertically and provides a safe and reliable measurement for children.
sprint performance | seven week intervention
  20 m Sprint: Electronic measurement of a timed (seconds) 20 m sprint, starting from a resting position. Start follows after an acoustic signal, with a precision of 1/100 second.
jump performance | seven week intervention
  Countermovement jump: Power per body mass, determined from a vertical countermovement jump (CMJ), has been shown to be correlated to leg extension strength in children while representing a more natural movement. The CMJ will be performed on a force plate (Leonardo Mechanograph®, Novotec medical, Pforzheim, Germany) with arms akimbo. The instruction will be to jump as high as possible. After familiarization, each participant performs 2-5 trials, with the best of the two trials with <5% difference being used for the analysis. The most important outcome parameter of this test is the maximum power output (peak power) normalized to body weight. The CMJ had a high intra-trial reproducibility (ICC>0.95) in 6-8 year old children, whereas inter-session variation has been reported to be high in children aged 6-12 years as well (ICC=0.95, SEE=1.92 standard error of estimate).
shuttle-run performance | seven week intervention
  20 m Shuttle-Run-test: This is a validated test which measures aerobic capacity by running forth and back for 20 m, with an initial running pace of 8.0 km/h and a progressive 0.5 km/every minute raise of the running speed given by a sound. The maximal performance will be reached when the child does not cross the 20 m line at the moment of the beep for two consecutive 20 m distances. Number of "paliers" (1 palier≅1 minute) performed will be counted with a precision of 0.5 paliers.
balance performance | seven week intervention
  This test of coordination includes balancing backward on 3 m long bars with a width of 3, 4.5, and 6 cm, respectively. The number of steps until the child's foot touches the floor will be counted; 3 trials will be performed for each bar width. The sum of these 9 tests will be used for statistical analysis.
object control | seven week intervention
  The Eye-Hand-Control test is valid and reliable and determines the level of controlling an object (tennis ball) while conducting repetitive movements (i.e., left-hand throw, right-hand catch, or right-hand throw, and left-hand catch, etc.) as frequently as possible in a time-constrained task of 30 sec. The children are free to use overhand and/or underhand techniques or a combination of both for throwing and catching. Children had to stand 1 m from a wall and throw the tennis ball at eye level on a wall. Participants conducted this test twice, with the number of successful ball catches across both trials resulting in the test score.
blood pressure, body composition | seven week intervention
  Anthropometry and blood pressure will be analysed on a seperate day, in a separate room parallel to the usual school lessons. 3 students will be evaluated at the same time.
side hop | seven week intervention
  Jumping sidewards: Measurement for speed and coordination. Jumping with both legs together on alternating sides of a bunton of wood, as many times as possible, within 15 seconds. Two trials will be performed. The number of jumps will be counted. The sum of the number of jumps of the two tests will be used for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport, Exercise and Health, Basel, Basellandschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No
No, because data is very sensible due to age of the participants.